CLINICAL TRIAL: NCT06271590
Title: The MAGICAL SV Trial - A Prospective, Multicenter, Randomized, Two-Arm, Single-blind Non Inferiority Trial to Evaluate the Safety and Efficacy of the MagicTouch™ Sirolimus-Coated Balloon in the Treatment of Small Vessels in Patients With Coronary Artery Disease.
Brief Title: MagicTouch™Sirolimus-Coated Balloon for Treatment of Coronary Artery Lesions in Small Vessels
Acronym: MAGICAL SV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concept Medical Inc. (Industry)
Collaborators: Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-US-R03
Record Dates: First submitted 2024-02-13; First posted 2024-02-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Native Coronary Artery Stenosis; Cardiovascular Diseases
Keywords: Drug coated balloon; Sirolimus coated balloon; De Novo; Magic Touch; SCB; Concept Medical; Small Vessel; MAGICAL SV
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases | interventions — Drug-Eluting Stents

STUDY DESIGN:
Intervention Model Description: 2:1 randomized trial (MagicTouchTM Sirolimus-Coated Balloon VS Drug eluting stent (ZES or EES)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- MagicTouch Sirolimus-Coated Balloon (SCB) (Experimental): Magic TouchTM is a Sirolimus Coated Balloon catheter intended to be used in coronary applications, treats the atherosclerosis of the coronary arteries by eluting the immunosuppressant agent Sirolimus without leaving behind a metallic scaffold.
  Interventions: Device: Sirolimus Drug Coated Balloon
- Drug eluting stents (DES) (Active Comparator): Everolimus eluting stents (EES) or Zotarolimus eluting stents (ZES)
  Interventions: Device: Drug eluting stents (DES)

INTERVENTIONS:
Device: Sirolimus Drug Coated Balloon — Magic TouchTM (Concept Medical) is a semi-compliant sirolimus drug coated balloon (SCB) for PCI, based on a polymer-free and nanocarrier based drug delivery technology.
  Other Names: Drug coated Balloon
  Arms: MagicTouch Sirolimus-Coated Balloon (SCB)
Device: Drug eluting stents (DES) — For subjects randomized to the control group (DES), the treating physician will choose an FDA cleared DES (ZES or EES) and follow lesion preparation and stent deployment according to the Instructions per use (IFU) and institutional practices.
  Arms: Drug eluting stents (DES)

SUMMARY:
This is a multicenter, randomized, single-blind pivotal study to evaluate the safety and efficacy of the MagicTouchTM Drug coated balloon in treatment of small vessels in patients with coronary artery disease. The objective is to establish the safety and efficacy of the Magic TouchTM Drug coated balloon in treatment of small vessels (≤2.75 mm).

A total of 1605 subjects will be enrolled in a maximum of 50 study sites located in North America. Additional sites located in Europe and South America may also participate in the study, with non-US sites contributing a maximum of ~50% of enrollees.

DETAILED DESCRIPTION:
Subjects with small vessel CAD (Coronary artery disease) presenting with lesions undergoing PCI (Percutaneous coronary intervention) will be randomized into two groups: treatment with the MagicTouch™ sirolimus-coated balloon or DCB (drug-coated balloon) on a 2:1 basis. Approximately 1605 subjects will be enrolled in the randomized study.

Treatment of a single lesion in a single major coronary artery or side branch will be enrolled per the inclusion and exclusion criteria. Target lesion must be located in a native coronary artery with a visually estimated diameter of<2.75 mm to length (including tandem lesions) ≤34.0 mm by visual estimation, and diameter stenosis ≥50% to <100% in symptomatic patients or ischemia by coronary physiology in patients without symptoms. The primary endpoint is TLF (target lesion failure) at 12 months after intervention.

All subjects providing informed consent will have their medical history reviewed and will undergo a physical examination, laboratory screen, and a standardized 12-lead ECG within 7 days of procedure. Women of childbearing potential will have a pregnancy test within one week prior to the procedure. SAQ-7 (Seattle Angina Questionnaire) will be collected at baseline, 30 days, 6 months, and 12 months and prior to any planned intervention.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Adult patient with an indication for PCI due to stable angina, NSTEACS, post-infarction angina or silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, FFR ≤0.80, or non-hyperemic pressure ratio [NHPR] ≤0.89 must be present)
2. Subject is ≥18 and <80 years old
3. Subject is willing to comply with all protocol-required follow-up evaluations and provides written informed consent

   Angiographic Inclusion Criteria:
4. Target reference vessel diameter (visual estimation) ≤2.75 mm
5. Successful lesion preparation (residual stenosis <30%), without flow-limiting complications (no or slow flow, dissection etc.)
6. Target lesion(s) in a native coronary artery
7. Up to two small vessel target lesions in two different vessels
8. Target lesion length (visual estimation): ≥6.0 and ≤34.0 mm and can be covered by a single 40 mm balloon
9. Target lesion diameter stenosis (visual estimation) >30% and <100% with Thrombolysis in Myocardial Infarction (TIMI) flow grade ≥2

Clinical Exclusion Criteria:

1. Planned (staged) intervention in the target vessel
2. ST-segment-elevation MI within 48 hours prior to index procedure
3. Subjects with acute cardiac decompensation or cardiogenic shock
4. Subject with a life expectancy of less than 24 months
5. Impaired renal function (glomerular filtration rate [GFR] <30 mL/min)
6. Documented left ventricular ejection fraction (LVEF) ≤30%
7. Known allergies to acetylsalicylic acid, clopidogrel, prasugrel, ticagrelor, heparin, contrast medium, sirolimus or similar drugs (i.e., ABT-578 [Zotarolimus], biolimus, tacrolimus)
8. Relative or absolute contraindication to dual antiplatelet therapy (DAPT) for at least 1 month (e.g., planned surgeries that cannot be delayed)
9. Subject has an indication for chronic oral anticoagulation treatment and a contraindication for concomitant treatment with a P2Y12 inhibitor
10. If femoral access is planned, significant peripheral arterial disease which precludes safe insertion of a 6F sheath
11. Hemoglobin <9 g/dL
12. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3
13. White blood cell count <3,000 cells/mm3
14. Active infection undergoing treatment
15. Clinically significant liver disease
16. Cerebrovascular accident (CVA) within 3 months or has any permanent neurological defect as a result of CVA
17. Subject is receiving oral or intravenous immunosuppressive therapy (e.g., inhaledsteroids are not excluded) or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus)
18. Subject is unlikely to comply with the follow up requirements, per investigator's assessment
19. Subject currently enrolled in other investigational device or drug trial in which primary endpoint has not been reached
20. Pregnant and/or breast-feeding females or females who intend to become pregnant during the time of the study

    Angiographic Exclusion Criteria:

    All exclusion criteria apply to the target lesion(s) or target vessel(s)
21. Re-stenotic lesion(s), whether due to percutaneous old balloon angioplasty (POBA) or prior stenting
22. True bifurcation lesion (lesion involves both main and side branch>2.5 mm) with planned treatment of both branches per investigator assessment
23. Angiographic evidence of thrombus in the target vessel
24. Myocardial bridging
25. Target lesion is heavily calcified
26. Diffuse distal disease to target lesion with impaired runoff, TIMI flow <2
27. Non-target lesion in the target vessel requiring PCI

Note: Non-target vessel PCI is allowed at the time of index procedure if performed prior to study intervention and if successful and uncomplicated. For target lesions located in branches of the three main vessels (left anterior descending artery [LAD], left circumflex artery [LCx], right coronary artery [RCA]), the term target vessel refers to the branch and not the main vessel.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1605 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure (TLF) | within 12 months
  the composite of cardiovascular mortality, target-vessel myocardial infarction (TV-MI) and ischemia driven target lesion revascularization

SECONDARY OUTCOMES:
Procedural success | at baseline, during the procedure
  defined as residual diameter stenosis <30% (DS), no flow-limiting dissection and with post-procedure The thrombolysis in myocardial infarction (TIMI) 3 flow, without the need for bailout stenting
Target lesion failure (TLF) | 30 days and at 6, 12, 24, 36, 48, and 60 months
  defined as the composite of cardiovascular mortality, target-vessel myocardial infarction (TVMI) and ischemia driven target lesion revascularization
Ischemia driven target vessel revascularization (ID-TVR) | 30 days and at 6, 12, 24, 36, 48, and 60 months
  Repeat revascularization of the target lesion due to recurrent ischemia
Target vessel revascularization (TVR) | 30 days and at 6, 12, 24, 36, 48, and 60 months
  Repeat revascularization of the target vessel
Any revascularization | 30 days and at 6, 12, 24, 36, 48, and 60 months
  any repeat PCI
Target vessel failure (TVF) | 30 days and at 6, 12, 24, 36, 48, and 60 months
  defined as the composite of cardiovascular mortality,ischemia driven TVR and TVMI
Q-wave myocardial infarction (MI) | 30 days and at 6, 12, 24, 36, 48, and 60 months
  Myocardial Infarction demonstrated by new pathological Q waves on ECG
Non Q-wave myocardial infarction (MI) | 30 days and at 6, 12, 24, 36, 48, and 60 months
  Myocardial Infarction not demonstrated by new pathological Q waves on ECG
Any myocardial infarction (MI) | 30 days and at 6, 12, 24, 36, 48, and 60 months
Target vessel myocardial infarction (TV MI) | 30 days and at 6, 12, 24, 36, 48, and 60 months
Spontaneous myocardial infarction (MI) | 30 days and at 6, 12, 24, 36, 48, and 60 months
Procedural myocardial infarction (MI) | Evaluated at 48 hours
Cardiovascular mortality | 30 days and at 6, 12, 24, 36, 48, and 60 months
All-cause mortality | 30 days and at 6, 12, 24, 36, 48, and 60 months
Cardiovascular mortality or myocardial infarction (MI) | 30 days and at 6, 12, 24, 36, 48, and 60 months
All-cause mortality or MI | 30 days and at 6, 12, 24, 36, 48, and 60 months
All-cause mortality, myocardial infarction (MI) or target vessel revascularization (TVR) | 30 days and at 6, 12, 24, 36, 48, and 60 months
Any probable or definite stent thrombosis | Evaluated at 48 hours
Probable stent thrombosis | 30 days and at 6, 12, 24, 36, 48, and 60 months
  Defined as per the Academic Research Consortium (ARC) criteria
Definite stent thrombosis | 30 days and at 6, 12, 24, 36, 48, and 60 months
  Defined as per the Academic Research Consortium (ARC) criteria

OTHER OUTCOMES:
Angina as assessed by SAQ-7 (Seattle Angina Questionnaire) | Quality of Life Endpoint evaluated at 30 days, 6 months, and 12 months
  Angina will be assessed at these specified timepoints and prior to any invasive procedure
  -Last angina assessment prior to any repeat coronary angiogram will be considered and subsequent assessments will be censored

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Dignity Health - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - University of Florida Health Sciences Center-Jacksonville, Jacksonville, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Tampa General Hospital / University of South Florida, Tampa, Florida
  - Emory University Hospital /Emory School of Medice, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Atlanticare Regional Medical Center, Pomona, New Jersey
  - University Hospitals, Cleveland Medical Center, Brooklyn, New York
  - North Shore University Hospital - Northwell, Manhasset, New York
  - Icahn School of Medicine at Mount Sinai/ Mount Sinai Hospital, New York, New York
  - Columbia University/NYP, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - University of Pittsburgh Medical center (UPMC), Pittsburgh, Pennsylvania
  - Baylor Scott & White The Heart Hospital - Plano, Plano, Texas
  - West Virginia University Heart & Vascular Institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No